CLINICAL TRIAL: NCT01731951
Title: A Pilot Open-Label Study of the Efficacy and Safety of Imetelstat (GRN163L) in Myelofibrosis and Other Myeloid Malignancies
Brief Title: Imetelstat Sodium in Treating Participants With Primary or Secondary Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR107110; CP14B019 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-11-18; First posted 2012-11-22 (Estimated); Results first posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-08

CONDITIONS: Primary Myelofibrosis; Secondary Myelofibrosis; Myeloid Malignancies
Keywords: Myelofibrosis; Myelodysplastic Syndromes; Myeloproliferative Neoplasm; Imetelstat; GRN163L
MeSH Terms: conditions — Primary Myelofibrosis; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — imetelstat; GRN163L peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A: Imetelstat 9.4 mg/kg (Myelofibrosis [MF]) (Experimental): Participants with MF regardless of spliceosome mutation status or presence of ring sideroblasts received imetelstat 9.4 milligram per kilogram (mg/kg), intravenously (IV) as 2-hour infusion on Day 1 of each 21-day cycle in Core Phase up to 9 cycles. Participants could receive imetelstat beyond Cycle 9 in the Extension Phase if they did not meet any of the withdrawal criteria, did not have disease progression and were receiving clinical benefit from treatment as determined by the investigator. Following treatment discontinuation, participants entered the Event Monitoring Phase for collection of survival status, disease status, and subsequent treatment information (Up to approximately 5.7 years).
  Interventions: Drug: Imetelstat
- Arm B: Imetelstat 9.4 mg/kg as Induction + Maintenance (MF) (Experimental): Participants with MF regardless of spliceosome mutation status or presence of ring sideroblasts received imetelstat 9.4 mg/kg, IV as 2-hour infusion on Days 1, 8, and 15 of 21-day cycle in Cycle 1 followed by 9.4 mg/kg on Day 1 of each 21-day cycle up to 9 cycles in the Core Phase. Participants could receive imetelstat beyond Cycle 9 in the Extension Phase if they did not meet any of the withdrawal criteria, did not have disease progression and were receiving clinical benefit from treatment as determined by the investigator. Following treatment discontinuation, participants entered the Event Monitoring Phase for collection of survival status, disease status, and subsequent treatment information (Up to approximately 5.7 years).
  Interventions: Drug: Imetelstat
- Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia) (Experimental): Participants with blast-phase myelofibrosis/acute myeloid leukemia (MF/AML) received imetelstat 9.4 mg/kg, IV as 2-hour infusion weekly on Days 1, 8, 15, 22 of a 28-day cycle up to 9 cycles in the Core Phase. Participants could receive imetelstat beyond Cycle 9 in the Extension Phase if they did not meet any of the withdrawal criteria, did not have disease progression and were receiving clinical benefit from treatment as determined by the investigator. Following treatment discontinuation, participants entered the Event Monitoring Phase for collection of survival status, disease status, and subsequent treatment information (Up to approximately 5.7 years).
  Interventions: Drug: Imetelstat
- Arm E: Imetelstat 7.5 - 9.4 mg/kg (MF [with Spliceosome Mutation or Ring Sideroblasts]) (Experimental): Participants with MF and spliceosome mutations or ring sideroblasts present received 2 cycles (Cycles 1-2) of imetelstat 7.5 mg/kg, IV as 2-hour infusion on Day 1 of a 28-day cycle followed by maintenance therapy with the same regimen or the possibility of dose escalation to imetelstat 9.4 mg/kg weekly if response to the initial dose was insufficient up to 9 cycles in the Core Phase. Participants could receive imetelstat beyond Cycle 9 in the Extension Phase if they did not meet any of the withdrawal criteria, did not have disease progression and were receiving clinical benefit from treatment as determined by the investigator. Following treatment discontinuation, participants entered the Event Monitoring Phase for collection of survival status, disease status, and subsequent treatment information (Up to approximately 5.7 years).
  Interventions: Drug: Imetelstat
- Arm F: Imetelstat 7.5 - 9.4 mg/kg (MF [without spliceosome mutation and ring sideroblasts]) (Experimental): Participants with MF without spliceosome mutations or ring sideroblasts present received 2 cycles (Cycles 1-2) of imetelstat 9.4 mg/kg, IV as 2-hour infusion on Day 1 of a 28-day cycle followed by maintenance therapy with the same regimen or imetelstat 7.5 mg/kg twice weekly on Days 1, 3 for 2 cycles of 28-day cycle (Cycles 3-4) followed by imetelstat 7.5 mg/kg 3-times-weekly on Days 1, 3, 5 of Cycles 5 and beyond of 28-day cycle up to 9 cycles in the Core Phase. Participants could receive imetelstat beyond Cycle 9 in the Extension Phase if they did not meet any of the withdrawal criteria, did not have disease progression and were receiving clinical benefit from treatment as determined by the investigator. Following treatment discontinuation, participants entered the Event Monitoring Phase for collection of survival status, disease status, and subsequent treatment information (Up to approximately 5.7 years).
  Interventions: Drug: Imetelstat
- Arm G: Imetelstat 7.5 - 9.4 mg/kg (MDS/MPN or MDS with Spliceosome Mutations or Ring Sideroblasts) (Experimental): Participants with either myelodysplastic syndromes/ myeloproliferative neoplasm (MDS/MPN) or MDS and spliceosome mutations or ring sideroblasts present received 2 cycles of 28-day cycle (Cycles 1-2) of imetelstat 7.5 mg/kg, IV as 2-hour infusion on Day 1 of a 28-day cycle followed by maintenance therapy with the same regimen or the possibility of dose escalation to imetelstat 9.4 mg/kg weekly if response to the initial dose was insufficient up to 9 cycles in the Core Phase. Participants could receive imetelstat beyond Cycle 9 in the Extension Phase if they did not meet any of the withdrawal criteria, did not have disease progression and were receiving clinical benefit from treatment as determined by the investigator. Following treatment discontinuation, participants entered the Event Monitoring Phase for collection of survival status, disease status, and subsequent treatment information (Up to approximately 5.7 years).
  Interventions: Drug: Imetelstat

INTERVENTIONS:
Drug: Imetelstat — Imetelstat sodium administered as IV over 2 hours with treatment as long as participants derive clinical benefit or until end of study.
  Other Names: GRN163L

SUMMARY:
This pilot clinical trial studies how well imetelstat sodium works in treating participants with primary or secondary myelofibrosis and other myeloid malignancies. Imetelstat sodium may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate overall response rate.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of imetelstat (imetelstat sodium) in myelofibrosis (MF).

II. To evaluate the efficacy of imetelstat in the reduction of spleen size, as measured by physical examination (palpable distance from the left costal margin).

III. To evaluate the efficacy of imetelstat in improving anemia or inducing red blood cell transfusion-independence in previously transfusion-dependent participants (per International Working Group for Myelofibrosis Research and Treatment [IWG-MRT] criteria).

IV. To evaluate onset and durability of response as defined in primary and secondary endpoints

EXPLORATORY OBJECTIVES:

I. To evaluate the effect of imetelstat on bone marrow histology, karyotype and JAK2V617F allele burden II. To evaluate the effect of imetelstat on leukocytosis, circulating blast count, circulating immature myeloid cell count and thrombocytosis.

OUTLINE: Participants receive imetelstat sodium intravenously (IV) over 2 hours on day 1. Participants may continue to receive imetelstat study treatment for as long as they derive clinical benefit or until study end. The study end when all participants discontinued study drug, the last participant enrolled has been treated for approximately 5.7 years, or imetelstat is commercially available in the United States, whichever occurs first.

Maximum duration of study was approximately 5.7 years. Arm C was never initiated, and participants allocated to Arm C (Imetelstat 9.4 mg/kg [with MF]) were reassigned to Arms A and B.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the following:
* Primary myelofibrosis (PMF) per the revised World Health Organization (WHO) criteria.
* Post-polycythemia vera/essential thrombocythemia myelofibrosis (Post-ET/PV MF) per the International Working Group for Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) criteria.
* High-risk or Intermediate-2 risk MF (as defined by the Dynamic International Prognostic Scoring System [DIPSS-plus]).
* Life expectancy of greater than or equal to (>=) 12 weeks.
* Able to provide informed consent and be willing to sign an informed consent form.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =<2.5 x upper limit of normal (ULN) (or =<5 x ULN if in the investigator's opinion the elevation is due to extramedullary hematopoiesis).
* Serum glutamic pyruvate transaminase (SGPT) alanine aminotransferase (ALT) =<2.5 x ULN (or =<5 x ULN if in the investigator's opinion the elevation is due to extramedullary hematopoiesis).
* Total bilirubin =<3.0 mg/dL (or direct bilirubin < 1 mg/dL).
* Creatinine =<3.0 mg/dL.
* Absolute neutrophil count >=1000/microliter (mcL).
* Platelet count >=50,000/mcL.
* Absence of active treatment with systemic anticoagulation and a baseline prothrombin time (PT) and activated partial thromboplastin time (aPTT) that does not exceed 1.5 x ULN.
* Females of childbearing potential must have a negative pregnancy test =<7 days prior to registration, unless they are surgically sterile for at least 3 months (i.e., hysterectomy), OR postmenopausal for at least 12 months (follicle-stimulating hormone [FSH] >30 U/mL).
* Females of childbearing potential must agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through end of study; permitted methods for preventing pregnancy must be communicated to study participants and their understanding confirmed.
* Males must agree to take appropriate precautions to avoid fathering a child (with at least 99% certainty) from screening through follow-up; permitted methods for preventing pregnancy should be communicated to the participants and their understanding confirmed.

Exclusion Criteria:

* Females who are pregnant or are currently breastfeeding.
* Any chemotherapy (e.g., hydroxyurea), immunomodulatory drug therapy (e.g., thalidomide), immunosuppressive therapy, corticosteroids > 10 mg/day prednisone or equivalent, growth factor treatment (e.g., erythropoietin) or Janus kinase (JAK) inhibitor therapy =<14 days prior to registration.
* Participants with another active malignancy.
* Note: participants with early stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin or cervical intraepithelial neoplasia are eligible for enrollment.
* Known positive status for human immunodeficiency virus (HIV).
* Any unresolved toxicity greater or equal to grade 2 from previous anticancer therapy, except for stable chronic toxicities not expected to resolve.
* Incomplete recovery from any prior surgical procedures or had surgery =<4 weeks prior to registration, excluding the placement of vascular access.
* Presence of acute active infection requiring antibiotics.
* Uncontrolled intercurrent illness or any concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the participant or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-10-29 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Clinical Team, Study Director — Geron Corporation
Locations (1):
- Rochester, Minnesota, United States

REFERENCES:
- [Derived] Tefferi A, Lasho TL, Begna KH, Patnaik MM, Zblewski DL, Finke CM, Laborde RR, Wassie E, Schimek L, Hanson CA, Gangat N, Wang X, Pardanani A. A Pilot Study of the Telomerase Inhibitor Imetelstat for Myelofibrosis. N Engl J Med. 2015 Sep 3;373(10):908-19. doi: 10.1056/NEJMoa1310523. PMID 26332545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1 site in the United States from 29 October 2012 to 22 January 2014 (end of recruitment). Data analyses includes data through 24 May 2018. Study has 4 phases: Screening Phase, Core Phase:up to nine 21-day (Arms A,B) or 28-day (Arms D,E,F,G) cycle, Extension Phase: after Cycle 9 to continue treatment with imetelstat; Event Monitoring Phase:Follow-up for those who discontinued treatment to collect survival status, disease status, and subsequent treatment information.
Pre-assignment Details: A total of 80 participants with Intermediate-2 or high-risk primary myelofibrosis (PMF)/post-polycythemia vera/essential thrombocythemia (post-PV/ET) MF (Arms A, B, C, E and F) or blast-phase MF (Arm D only) or spliceosome-mutated (or with ring sideroblasts) myelodysplastic syndromes [MDS]/ myeloproliferative neoplasm [MPN] (Arm G only) were enrolled to receive imetelstat. Arm C (Imetelstat 9.4 mg/kg [with MF]) was never initiated, participants allocated to Arm C were reassigned to Arm A or B.
Groups:
- Arm A: Imetelstat 9.4 mg/kg (MF): Participants with MF regardless of spliceosome mutation status or presence of ring sideroblasts received imetelstat 9.4 milligram per kilogram (mg/kg), intravenously (IV) as 2-hour infusion on Day 1 of each 21-day cycle in Core Phase up to 9 cycles. Participants could receive imetelstat beyond Cycle 9 in the Extension Phase if they did not meet any of the withdrawal criteria, did not have disease progression and were receiving clinical benefit from treatment as determined by the investigator. Following treatment discontinuation, participants entered the Event Monitoring Phase for collection of survival status, disease status, and subsequent treatment information (Up to approximately 5.7 years).
Period: Overall Study
Arm/Group | Arm A: Imetelstat 9.4 mg/kg (MF) | Arm B: Imetelstat 9.4 mg/kg as Induction + Maintenance (MF) | Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia) | Arm E: Imetelstat 7.5 - 9.4 mg/kg (MF [With Spliceosome Mutation or Ring Sideroblasts]) | Arm F: Imetelstat 7.5 - 9.4 mg/kg (MF [Without Spliceosome Mutation and Ring Sideroblasts]) | Arm G: Imetelstat 7.5 - 9.4 mg/kg (MDS/MPN or MDS With Spliceosome Mutations or Ring Sideroblasts)
Started | 19 | 16 | 9 | 9 | 18 | 9
Completed | 2 | 1 | 0 | 0 | 6 | 0
Not Completed | 17 | 15 | 9 | 9 | 12 | 9
Not completed — Documented Disease Progression | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 1 | 3 | 1
Not completed — Withdrawal of Consent | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 13 | 15 | 9 | 8 | 9 | 6

BASELINE CHARACTERISTICS:
Population: All Treated Analysis Set included all participants who received at least one dose of imetelstat.
Groups:
- Arm A: Imetelstat 9.4 mg/kg (MF): Participants with MF regardless of spliceosome mutation status or presence of ring sideroblasts received imetelstat 9.4 mg/kg, IV as 2-hour infusion on Day 1 of each 21-day cycle in Core Phase up to 9 cycles. Participants could receive imetelstat beyond Cycle 9 in the Extension Phase if they did not meet any of the withdrawal criteria, did not have disease progression and were receiving clinical benefit from treatment as determined by the investigator. Following treatment discontinuation, participants entered the Event Monitoring Phase for collection of survival status, disease status, and subsequent treatment information (Up to approximately 5.7 years).
- Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia): Participants with blast-phase MF/AML received imetelstat 9.4 mg/kg, IV as 2-hour infusion weekly on Days 1, 8, 15, 22 of a 28-day cycle up to 9 cycles in the Core Phase. Participants could receive imetelstat beyond Cycle 9 in the Extension Phase if they did not meet any of the withdrawal criteria, did not have disease progression and were receiving clinical benefit from treatment as determined by the investigator. Following treatment discontinuation, participants entered the Event Monitoring Phase for collection of survival status, disease status, and subsequent treatment information (Up to approximately 5.7 years).
- Arm G: Imetelstat 7.5 - 9.4 mg/kg (MDS/MPN or MDS With Spliceosome Mutations or Ring Sideroblasts): Participants with either MDS/MPN or MDS and spliceosome mutations or ring sideroblasts present received 2 cycles of 28-day cycle (Cycles 1-2) of imetelstat 7.5 mg/kg, IV as 2-hour infusion on Day 1 of a 28-day cycle followed by maintenance therapy with the same regimen or the possibility of dose escalation to imetelstat 9.4 mg/kg weekly if response to the initial dose was insufficient up to 9 cycles in the Core Phase. Participants could receive imetelstat beyond Cycle 9 in the Extension Phase if they did not meet any of the withdrawal criteria, did not have disease progression and were receiving clinical benefit from treatment as determined by the investigator. Following treatment discontinuation, participants entered the Event Monitoring Phase for collection of survival status, disease status, and subsequent treatment information (Up to approximately 5.7 years).
- Total: Total of all reporting groups
Arm/Group | Arm A: Imetelstat 9.4 mg/kg (MF) | Arm B: Imetelstat 9.4 mg/kg as Induction + Maintenance (MF) | Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia) | Arm E: Imetelstat 7.5 - 9.4 mg/kg (MF [With Spliceosome Mutation or Ring Sideroblasts]) | Arm F: Imetelstat 7.5 - 9.4 mg/kg (MF [Without Spliceosome Mutation and Ring Sideroblasts]) | Arm G: Imetelstat 7.5 - 9.4 mg/kg (MDS/MPN or MDS With Spliceosome Mutations or Ring Sideroblasts) | Total
Number analyzed (Participants) | 19 | 16 | 9 | 9 | 18 | 9 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 6 | 1 | 10 | 3 | 35
  >=65 years | 11 | 9 | 3 | 8 | 8 | 6 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 3 | 3 | 7 | 2 | 26
  Male | 12 | 12 | 6 | 6 | 11 | 7 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 15 | 8 | 9 | 17 | 7 | 75
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 1 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 19 | 15 | 6 | 9 | 17 | 8 | 74
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 1 | 1 | 4
Eastern Cooperative Oncology Group (ECOG) Performance Status Score [Count of Participants; unit: Participants] — ECOG Performance Status has 5 Scores.0= Fully active, able to carry on all predisease performance without restriction;1= Restricted in physically strenuous activity but ambulatory and able to carry out work on a light/sedentary nature,2= Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours;3= Capable of only limited self-care; confined to bed/chair more than 50% of waking hours;4= Completely disabled. Cannot carry on any self-care.Totally confined to bed/chair;5= Dead. Number of participants for each score are reported.
  Participants
    0 | 7 | 5 | 2 | 1 | 2 | 2 | 19
    1 | 11 | 6 | 4 | 4 | 13 | 7 | 45
    2 | 1 | 5 | 3 | 4 | 3 | 0 | 16
    3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelofibrosis subtype [Count of Participants; unit: Participants] — Myelofibrosis subtypes included MDS/MPN or MDS, blast-phase myelofibrosis, primary myelofibrosis, post-ET myelofibrosis, and Post-PV myelofibrosis. Number of participants for each subtype are reported.
  Participants
    Myelodysplastic Syndromes/ Myeloproliferative Neoplasm (MDS/MPN) or MDS | 0 | 0 | 0 | 0 | 0 | 9 | 9
    Blast-phase Myelofibrosis | 0 | 0 | 8 | 0 | 0 | 0 | 8
    Primary Myelofibrosis | 11 | 8 | 0 | 7 | 9 | 0 | 35
    Post-Essential Thrombocythemia (ET) Myelofibrosis | 1 | 5 | 1 | 2 | 5 | 0 | 14
    Post-Polycythemia Vera (PV) Myelofibrosis | 7 | 3 | 0 | 0 | 4 | 0 | 14
Dynamic International Prognostic Scoring System (DIPSS)-Plus Risk Status [Count of Participants; unit: Participants] — DIPSS stratifies primary myelofibrosis (PMF) into four risk categories (low, intermediate 1, intermediate 2, and high risk), based on 5 clinical factors; Age>65, Hemoglobin <10 grams per deciliter (gm/dL), Leukocytes >10 (9)/L, circulating blasts ≥1%, and constitutional symptoms. Participants for each status are reported. Only categories with data are reported. Population: Number analyzed is the number of participants with data available for DIPSS-Plus risk status.
  Participants
    number analyzed (Participants) | 19 | 16 | 9 | 9 | 18 | 8 | 79
    Intermediate-2 Risk (2 or 3 risk factors) | 11 | 5 | 1 | 1 | 10 | 6 | 34
    High Risk (4 or more risk factors) | 8 | 11 | 8 | 8 | 8 | 2 | 45
Spliceosomal Mutation Status [Count of Participants; unit: Participants] — Spliceosome mutations represent a group of acquired genetic alterations that affect both myeloid and lymphoid malignancies. Population: Number analyzed is the number of participants with data available for spliceosomal mutation status.
  Participants
    number analyzed (Participants) | 19 | 15 | 7 | 9 | 18 | 9 | 77
    Had Spliceosomal Mutation | 7 | 4 | 5 | 8 | 0 | 7 | 31
    Had No Spliceosomal Mutation | 12 | 11 | 2 | 1 | 18 | 2 | 46
Spliceosomal Mutation Type [Count of Participants; unit: Participants] — Spliceosome mutations represent a group of acquired genetic alterations that affect both myeloid and lymphoid malignancies. Spliceosomal mutation type included SF3B1, SRSF2 and U2AF1. Number of participants for each type are reported. Population: Number analyzed is the number of participants with data available for spliceosomal mutation type.
  Participants
    number analyzed (Participants) | 7 | 4 | 5 | 8 | 0 | 7 | 31
    Splicing Factor 3B Subunit 1 (SF3B1) | 1 | 2 | 1 | 1 |  | 6 | 11
    Serine And Arginine Rich Splicing Factor 2 (SRSF2) | 2 | 1 | 2 | 4 |  | 0 | 9
    U2 Small Nuclear RNA Auxiliary Factor 1 (U2AF1) | 4 | 1 | 2 | 3 |  | 1 | 11
Ringed Sideroblasts Present [Count of Participants; unit: Participants] — Ring sideroblasts are erythroblasts with iron-loaded mitochondria visualized by Prussian blue staining (Perls' reaction) as a perinuclear ring of blue granules. Refractory anemia with ring sideroblasts (RARS) is a type of MDS that is characterized by anemia and the presence of at least 15 percent ring sideroblasts in the marrow. Population: Number analyzed is the number of participants with data available for ringed sideroblasts present.
  Participants
    number analyzed (Participants) | 16 | 12 | 6 | 9 | 17 | 9 | 69
    Yes | 4 | 2 | 1 | 3 | 0 | 8 | 18
    No | 12 | 10 | 5 | 6 | 17 | 1 | 51
JAK2V617F Mutation [Count of Participants; unit: Participants] — JAK2 V617F mutation is an acquired, somatic mutation present in the majority of participants with myeloproliferative cancer (myeloproliferative neoplasms) i.e. nearly 100% of participants with polycythemia vera and in about 50% of participants with essential thrombocytosis and primary myelofibrosis. Population: Number analyzed is the number of participants with data available for JAK2V617F Mutation.
  Participants
    number analyzed (Participants) | 16 | 14 | 9 | 9 | 18 | 9 | 75
    Had JAK2V617F Mutation | 15 | 8 | 5 | 6 | 14 | 3 | 51
    Had No JAK2V617F Mutation | 1 | 5 | 4 | 3 | 4 | 6 | 23
    Unable to Determine | 0 | 1 | 0 | 0 | 0 | 0 | 1
Transfusion Dependent [Count of Participants; unit: Participants] — Transfusion dependency was defined by a history of at least 2 units of red blood cell transfusions in the last month for a hemoglobin level of less than 85 grams per deciliter (g/dL) that was not associated with clinically overt bleeding.
  Participants
    Had Transfusion Dependency | 8 | 5 | 3 | 2 | 4 | 5 | 27
    Had No Transfusion Dependency | 11 | 11 | 6 | 7 | 14 | 4 | 53

OUTCOME MEASURES:

1. Primary Outcome: MF Participants: Percentage of Participants With Overall Response (OR) - (Clinical Improvement[CI] or Partial Remission[PR] or Complete Remission[CR]) Per International Working Group - Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) Criteria
Description: OR:CI/PR/CR per IWG-MRT. CR:Bone marrow (BM):<5% blasts;≤Grade 1 MF, AND Peripheral blood:Hemoglobin (Hb) ≥100 g/liter (g/L) and <upper normal limit (UNL);Neutrophil count(NC) ≥1x10^9/L and <UNL; Platelet(PLT) count ≥100x10^9/L and <UNL;<2% immature myeloid cells(IMCs), AND Clinical: Resolution of disease symptoms; Spleen and liver not palpable; No evidence of extramedullary hematopoeisis(EMH). PR:All CR criteria plus peripheral blood: Hb≥85 but <100g/L and <UNL; NC ≥1x10^9/L and <UNL; PLT count ≥50 but <100x10^9/L and <UNL;<2%IMCs. CI:achievement of anemia (≥20 g/L increase in Hb level), spleen(baseline splenomegaly palpable at 5-10 cm, below left costal margin(LCM), becomes not palpable), symptoms response (50% reduction in total symptom score) without progressive disease (PD) (appearance of new splenomegaly- palpable at least [≥]5 cm below LCM)/increase in severity of anemia, thrombocytopenia/neutropenia. Data is reported separately for arms whose response was assessed per IWG-MRT.
Time Frame: Up to first 9 cycles of treatment (each cycle was of 21 days for Arms A and B and 28 days for Arms E and F)
Population: Eligible Analysis Set included subset of all participants who received at least one dose of study drug that excludes ineligible participants who did not satisfy each and every eligibility criteria for study entry. Data is reported for arm groups (Arms A, B, E and F) whose overall response was assessed by IWG-MRT criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Imetelstat 9.4 mg/kg (MF) | Arm B: Imetelstat 9.4 mg/kg as Induction + Maintenance (MF) | Arm E: Imetelstat 7.5 - 9.4 mg/kg (MF [With Spliceosome Mutation or Ring Sideroblasts]) | Arm F: Imetelstat 7.5 - 9.4 mg/kg (MF [Without Spliceosome Mutation and Ring Sideroblasts])
Number analyzed (Participants) | 19 | 14 | 9 | 18
percentage of participants | 36.84 [15.2 to 58.5] | 35.7 [10.6 to 60.8] | 0 [NA to NA] — Upper and lower limits of 95% CI were not estimable due to limited number of participants with the event. | 33.3 [11.6 to 55.1]

2. Primary Outcome: Blastic MF/AML Participants: Percentage of Participants With Overall Response
Description: For this pilot study, overall response was defined as achievement of a leukemic response (i.e. a clinically meaningful reduction in Blast cells). This was quantified as <5% peripheral blood and bone marrow blasts % that lasts for at least two months. Data is reported separately for this arm where response was assessed by this specific criterion.
Time Frame: Up to first 9 cycles of treatment (each cycle was of 28 days for Arm D)
Population: All Treated Analysis Set included all participants who received at least one dose of study drug. Data is reported for Arm D: Imetelstat 9.4 mg/kg (Blastic MF/AML) participants whose overall response was assessed by a specific criterion.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia)
Number analyzed (Participants) | 9
percentage of participants | 0 [NA to NA] — Upper and lower limits of 95% CI were not estimable due to limited number of participants with the event.

3. Primary Outcome: MDS Participants: Percentage of Participants With Overall Response (Hematologic Improvement [HI] or PR or CR) Per IWG Criteria
Description: OR: HI/PR/CR per IWG. CR: BM:≤5% myeloblasts (all cell lines normal maturation), Peripheral blood:Hgb ≥11g/dL, PLTs ≥100x10^9/L, Neutrophils ≥1.0x10^9/L, Blasts 0%. PR: All CR criteria if abnormal before treatment except- BM blasts decreased ≥50% over pretreatment but still >5%, Cellularity, morphology not relevant. HI responses:1) Erythroid: Hgb increase ≥1.5 g/dL, Relevant reduction of red blood cell(RBC) units transfusions by absolute ≥4 RBC transfusions/8 week (wk) compared with pretreatment transfusion number in previous 8 wk. Only RBC transfusions given for Hgb of ≤9.0 g/dL.2)PLTs:Absolute increase ≥30x10^9/L starting >20x10^9/L PLTs; Increase from <20x10^9/L to >20x10^9/L and by ≥100%; 3)Neutrophil: ≥100% increase, absolute increase >0.5x10^9/L; 4)Progression/relapse after HI:≥1 of following:≥50% decrement from maximum response levels in granulocytes/PLTs, Reduction in Hgb ≥1.5 g/dL,Transfusion dependence. Data is reported separately for arm whose response was assessed per IWG.
Time Frame: Up to first 9 cycles of treatment (each cycle was of 28 days for Arm G)
Population: All Treated Analysis Set included all participants who received at least one dose of the study drug. Data is reported for Arm G: Imetelstat 9.4 mg/kg (MDS/MPN or MDS and spliceosome mutations or ring sideroblasts) participants whose overall response was assessed by IWG criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm G: Imetelstat 7.5 - 9.4 mg/kg (MDS/MPN or MDS With Spliceosome Mutations or Ring Sideroblasts)
Number analyzed (Participants) | 9
percentage of participants | 33.3 [2.5 to 64.1]

4. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs), Grade >= 3 TEAEs and Treatment Related Adverse Events
Description: TEAEs defined as those events that 1) occur on or after the first dose of study drug, through the treatment phase, and for 30 days following the last dose of study drug or until subsequent anti-cancer therapy if earlier; 2) any event that is considered study drug-related regardless of the start date of the event; or 3) any event that is present at baseline but worsens in severity or is subsequently considered drug-related by the investigator. Grade >=3 TEAE defined as events that are severe, life-threatening or disabling, or fatal and considered related to imetelstat as per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. An AE was considered related to the study drug if the event was assessed by the investigator as probably or possibly related.
Time Frame: From first dose of study drug up to 30 days from the last dose of study drug or until subsequent anti-cancer therapy if earlier (Up to approximately 5.7 years)
Population: All Treated Analysis Set included all participants who received at least one dose of imetelstat.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Imetelstat 9.4 mg/kg (MF) | Arm B: Imetelstat 9.4 mg/kg as Induction + Maintenance (MF) | Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia) | Arm E: Imetelstat 7.5 - 9.4 mg/kg (MF [With Spliceosome Mutation or Ring Sideroblasts]) | Arm F: Imetelstat 7.5 - 9.4 mg/kg (MF [Without Spliceosome Mutation and Ring Sideroblasts]) | Arm G: Imetelstat 7.5 - 9.4 mg/kg (MDS/MPN or MDS With Spliceosome Mutations or Ring Sideroblasts)
Number analyzed (Participants) | 19 | 16 | 9 | 9 | 18 | 9
percentage of participants
  TEAEs | 100 | 100 | 100 | 100 | 100 | 100
  Grade >=3 TEAEs | 100 | 93.5 | 100 | 77.8 | 83.3 | 100
  Treatment Related AEs | 89.5 | 75 | 88.9 | 77.8 | 83.3 | 100

5. Secondary Outcome: Number of Participants With Spleen Response Per IWG-MRT Criteria
Description: Spleen response per IWG-MRT criteria defined as baseline splenomegaly that is palpable at 5-10 cm, below the LCM, becomes not palpable, OR A baseline splenomegaly that is palpable at >10 cm, below the LCM, decreases by ≥50%. Baseline splenomegaly that is palpable at <5 cm, below the LCM, is not eligible for spleen response. Confirmation by Magnetic resonance imaging (MRI) or computerized tomography (CT) showing ≥35% spleen volume reduction is recommended (but not required). Spleen response was assessed only in participants with MF.
Time Frame: Up to approximately 5.7 years
Population: Arms A, B, E and F: Eligible Analysis Set included subset of all participants who received at least one dose of study drug that excludes ineligible participants who did not satisfy each and every eligibility criteria for study entry. Arm D: All Treated Analysis Set included all participants who received at least one dose of imetelstat.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Imetelstat 9.4 mg/kg (MF) | Arm B: Imetelstat 9.4 mg/kg as Induction + Maintenance (MF) | Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia) | Arm E: Imetelstat 7.5 - 9.4 mg/kg (MF [With Spliceosome Mutation or Ring Sideroblasts]) | Arm F: Imetelstat 7.5 - 9.4 mg/kg (MF [Without Spliceosome Mutation and Ring Sideroblasts])
Number analyzed (Participants) | 19 | 14 | 9 | 9 | 18
Participants | 3 | 1 | 1 | 0 | 2

6. Secondary Outcome: MF and Blastic MF/AML Participants: Number of Participants With Transfusion Independence (CI by Anemia Response) Per IWG-MRT
Description: Transfusion dependency was defined by a history of at least 2 units of red blood cell transfusions in the last month for a hemoglobin level of less than 85 g/L that was not associated with clinically overt bleeding. A participant who was transfusion dependent at baseline was considered transfusion independent if the participant met either of the following conditions: Received no more than 1 unit of red blood cell transfusions in a rolling time interval of 30 days or more, and had a hemoglobin level increase over baseline more than 2 g/dL if participant baseline hemoglobin level was less than 85 g/L and received no transfusion. Anemia response per IWG-MRT Criteria- Transfusion-independent participants: a ≥20 g/L increase in hemoglobin level. Transfusion-dependent participants: becoming transfusion-independent. Data is reported separately for arms assessed as per the IWG-MRT criteria.
Time Frame: Up to approximately 5.7 years
Population: Arms A, B, E, F: Eligible Analysis Set included subset of all participants who received at least one dose of study drug that excludes ineligible participants who did not satisfy each and every eligibility criteria for study entry. Arm D: All Treated Analysis Set included all participants who received at least one dose of imetelstat, assessed per IWG-MRT.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Imetelstat 9.4 mg/kg (MF) | Arm B: Imetelstat 9.4 mg/kg as Induction + Maintenance (MF) | Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia) | Arm E: Imetelstat 7.5 - 9.4 mg/kg (MF [With Spliceosome Mutation or Ring Sideroblasts]) | Arm F: Imetelstat 7.5 - 9.4 mg/kg (MF [Without Spliceosome Mutation and Ring Sideroblasts])
Number analyzed (Participants) | 19 | 14 | 9 | 9 | 18
Participants | 1 | 0 | 0 | 0 | 3

7. Secondary Outcome: MDS Participants: Number of Participants With Transfusion Independence (HI by Erythroid Response) Per IWG Criteria
Description: Transfusion dependency was defined by a history of at least 2 units of red blood cell transfusions in the last month for a hemoglobin level of less than 85 g/L that was not associated with clinically overt bleeding. A participant who was transfusion dependent at baseline was considered transfusion independent if the participant met either of the following conditions: Received no more than 1 unit of red blood cell transfusions in a rolling time interval of 30 days or more, and had a hemoglobin level increase over baseline more than 2 g/dL if participant baseline hemoglobin level was less than 85 g/L and received no transfusion. HI responses included: 1) Erythroid: Hgb increase ≥1.5 g/dL, Relevant reduction of RBC units transfusions by absolute number of >=4 RBC transfusions/8 week compared with pretreatment transfusion number in previous 8 week. Only RBC transfusions given for Hgb of ≤9.0 g/dL. Data is reported separately for arm assessed as per IWG criteria.
Time Frame: Up to approximately 5.7 years
Population: All Treated Analysis Set included all participants who received at least one dose of study drug. Data is reported for Arm G: Imetelstat 9.4 mg/kg (MDS/MPN or MDS and spliceosome mutations or ring sideroblasts) participants whose transfusion independence (HI by erythroid response) was assessed by IWG criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm G: Imetelstat 7.5 - 9.4 mg/kg (MDS/MPN or MDS With Spliceosome Mutations or Ring Sideroblasts)
Number analyzed (Participants) | 9
Participants | 3

8. Secondary Outcome: MF Participants: Time to Response
Description: Time to response was defined as the duration from study Day 1 to the earliest date that a response is first documented. The response CI/CR/PR was assessed by IWG-MRT criteria.
Time Frame: From study Day 1 to the earliest date that a response was first documented (Up to approximately 5.7 years)
Population: Eligible Analysis Set included subset of all participants who received at least one dose of study drug that excludes ineligible participants who did not satisfy each and every eligibility criteria for study entry. Data is reported for arm groups (Arms A, B, E and F) whose overall response was assessed by IWG-MRT criteria. Only responders were analyzed for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Imetelstat 9.4 mg/kg (MF) | Arm B: Imetelstat 9.4 mg/kg as Induction + Maintenance (MF) | Arm E: Imetelstat 7.5 - 9.4 mg/kg (MF [With Spliceosome Mutation or Ring Sideroblasts]) | Arm F: Imetelstat 7.5 - 9.4 mg/kg (MF [Without Spliceosome Mutation and Ring Sideroblasts])
Number analyzed (Participants) | 7 | 5 | 0 | 6
months | 2.1 [0.7 to 3.5] | 1.4 [0.7 to 5.6] |  | 2.9 [1.9 to 12.1]

9. Secondary Outcome: Blastic MF/AML Participants: Time to Response
Description: Time to response was defined as the duration from study Day 1 to the earliest date that a response is first documented. Response was defined as achievement of a leukemic response (i.e. a clinically meaningful reduction in Blast cells). This was quantified as <5% peripheral blood and bone marrow blasts % that lasts for at least two months. Data for time to response is reported as per criteria of response assessment.
Time Frame: From study Day 1 to the earliest date that a response was first documented (Up to approximately 5.7 years)
Population: All Treated Analysis Set included all participants who received at least one dose of the study drug. Only responders were analyzed for this outcome measure. Data is reported for Arm D: Imetelstat 9.4 mg/kg (Blastic MF/AML) participants whose overall response was assessed by a specific criterion.
Arm/Group | Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia)
Number analyzed (Participants) | 0

10. Secondary Outcome: MDS Participants: Time to Response
Description: Time to response was defined as the duration from study Day 1 to the earliest date that a response is first documented. Response was defined as HI, PR or CR per IWG criteria. Data for time to response is reported as per criteria of response assessment.
Time Frame: From study Day 1 to the earliest date that a response was first documented (Up to approximately 5.7 years)
Population: All Treated Analysis Set included all participants who received at least one dose of the study drug. Only responders were analyzed for this outcome measure. Data is reported for Arm G: Imetelstat 9.4 mg/kg (MDS/MPN or MDS and spliceosome mutations or ring sideroblasts) participants whose overall response was assessed by IWG criteria.
Measure: Median (Full Range); unit: months
Arm/Group | Arm G: Imetelstat 7.5 - 9.4 mg/kg (MDS/MPN or MDS With Spliceosome Mutations or Ring Sideroblasts)
Number analyzed (Participants) | 3
months | 3.7 [2.8 to 4.9]

11. Secondary Outcome: MF Participants: Duration of Response (DOR) Per IWG-MRT Criteria
Description: DOR measured from time of initial response (CR/PR/CI) until documented PD or death whichever occurs first. If no PD/death occurs DOR is censored at last disease evaluation date for responders. CR:BM: <5%blasts; ≤Grade 1 MF, AND Peripheral blood:Hb≥100 g/L and <UNL;Neutrophil count≥1x10^9/L and <UNL;PLT count≥100x10^9/L and <UNL;<2% IMCs, AND Clinical:Resolution of disease symptoms;Spleen and liver not palpable;No evidence of EMH.PR:All CR criteria plus peripheral blood:Hb≥85 but <100g/L and <UNL;NC≥1x10^9/L and <UNL;PLTcount ≥50 but<100x10^9/L and<UNL;<2%IMCs. CI:achievement of anemia(≥20 g/L increase Hb level),spleen(baseline splenomegaly-palpable at 5-10cm,below LCM,becomes not palpable) or symptoms response(50% reduction in total symptom score) without PD(appearance of new splenomegaly- palpable[>= 5 cm below LCM) or increase in severity of anemia, thrombocytopenia or neutropenia. Data is reported separately for arms whose DOR was assessed per IWG-MRT. Kaplan-Meier method was used.
Time Frame: From time of initial response until documented disease progression or death whichever occurs first (Up to approximately 5.7 years)
Population: Eligible Analysis Set included subset of all participants who received at least one dose of study drug that excludes ineligible participants who did not satisfy each and every eligibility criteria for study entry. Data is reported for arm groups whose DOR was assessed by IWG-MRT criteria. Only responders were analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Imetelstat 9.4 mg/kg (MF) | Arm B: Imetelstat 9.4 mg/kg as Induction + Maintenance (MF) | Arm E: Imetelstat 7.5 - 9.4 mg/kg (MF [With Spliceosome Mutation or Ring Sideroblasts]) | Arm F: Imetelstat 7.5 - 9.4 mg/kg (MF [Without Spliceosome Mutation and Ring Sideroblasts])
Number analyzed (Participants) | 7 | 5 | 0 | 6
months | 24.36 [17.94 to 40.74] | NA [16.59 to NA] — Median and upper limit of 95% CI were not estimable due to limited number of participants with the event. |  | 35.52 [NA to NA] — Upper and lower limits of 95% CI were not estimable due to limited number of participants with the event.

12. Secondary Outcome: Blastic MF/AML Participants: Duration of Response
Description: DOR was measured from the time of initial response until documented disease progression or death whichever occurs first. If no PD/death occurs the DOR is censored at last disease evaluation date for responders. Response is defined as achievement of <5% peripheral blood and bone marrow blast % that lasts for at least two months. PD is the appearance of new splenomegaly that is palpable at least 5 cm below the LCM. Data is reported separately for arm whose DOR was assessed by a specific criterion. Kaplan-Meier method was used.
Time Frame: as for outcome 11
Population: All Treated Analysis Set included all participants who received at least one dose of the study drug. Data is reported for Arm D: Imetelstat 9.4 mg/kg (Blastic MF/AML) participants whose DOR was assessed by a specific criterion. Only responders were analyzed for this outcome measure.
Arm/Group | Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia)
Number analyzed (Participants) | 0

13. Secondary Outcome: MDS Participants: Duration of Response Per IWG Criteria
Description: DOR: time of initial response (CR/PR/HI) until documented PD/death whichever occurs first. If no PD/death occurs DOR is censored at last disease evaluation date for responders. Data reported separately for arm assessed per IWG. Kaplan-Meier method was used.
Time Frame: From the time of initial response (CR/PR/HI) until documented disease progression or death whichever occurs first (Up to approximately 5.7 years)
Population: All Treated Analysis Set included all participants who received at least one dose of the study drug. Data is reported for Arm G: Imetelstat 9.4 mg/kg (MDS/MPN or MDS and spliceosome mutations or ring sideroblasts) participants whose DOR was assessed by IWG criteria. Only responders were analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm G: Imetelstat 7.5 - 9.4 mg/kg (MDS/MPN or MDS With Spliceosome Mutations or Ring Sideroblasts)
Number analyzed (Participants) | 3
months | NA [NA to NA] — Median, upper and lower limits of 95% CI were not estimable as all DOR of responder participants were censored .

14. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the as the interval from Study Day 1 to the date of death from any cause. Survival time of living participants was censored on the last date a participant is known to be alive or lost to follow-up. Overall Survival was estimated by Kaplan-Meier method.
Time Frame: From Study Day 1 to the date of death from any cause (Up to approximately 5.7 years)
Population: All Treated Analysis Set included all participants who received at least one dose of imetelstat.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Imetelstat 9.4 mg/kg (MF) | Arm B: Imetelstat 9.4 mg/kg as Induction + Maintenance (MF) | Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia) | Arm E: Imetelstat 7.5 - 9.4 mg/kg (MF [With Spliceosome Mutation or Ring Sideroblasts]) | Arm F: Imetelstat 7.5 - 9.4 mg/kg (MF [Without Spliceosome Mutation and Ring Sideroblasts]) | Arm G: Imetelstat 7.5 - 9.4 mg/kg (MDS/MPN or MDS With Spliceosome Mutations or Ring Sideroblasts)
Number analyzed (Participants) | 19 | 16 | 9 | 9 | 18 | 9
months | 42.61 [19.12 to 56.77] | 26.73 [16.46 to 36.17] | 4.93 [1.05 to 15.67] | 12.09 [7.06 to 27.14] | NA [12.22 to NA] — Median and upper limit of 95% CI were not estimable due to limited number of participants with the event. | 28.42 [6.64 to NA] — Upper limit of 95% CI was not estimable due to limited number of participants with the event.

ADVERSE EVENTS:
Time Frame: From first dose of study drug to the last dose of study drug or until subsequent anti-cancer therapy if earlier (Up to approximately 5.7 years)
Description: All treated analysis set included all participants who received at least 1 dose of Imetelstat. All non-serious adverse events (at 5% threshold) and serious adverse event including requirements for expedited reporting of serious adverse events occurring within 30 days of the last dose of study drug are reported.
Groups:
- Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia: Participants with blast-phase MF/AML received imetelstat 9.4 mg/kg, IV as 2-hour infusion weekly on Days 1, 8, 15, 22 of a 28-day cycle up to 9 cycles in the Core Phase. Participants could receive imetelstat beyond Cycle 9 in the Extension Phase if they did not meet any of the withdrawal criteria, did not have disease progression and were receiving clinical benefit from treatment as determined by the investigator. Following treatment discontinuation, participants entered the Event Monitoring Phase for collection of survival status, disease status, and subsequent treatment information (Up to approximately 5.7 years).
Arm/Group | Arm A: Imetelstat 9.4 mg/kg (MF) | Arm B: Imetelstat 9.4 mg/kg as Induction + Maintenance (MF) | Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia | Arm E: Imetelstat 7.5 - 9.4 mg/kg (MF [With Spliceosome Mutation or Ring Sideroblasts]) | Arm F: Imetelstat 7.5 - 9.4 mg/kg (MF [Without Spliceosome Mutation and Ring Sideroblasts]) | Arm G: Imetelstat 7.5 - 9.4 mg/kg (MDS/MPN or MDS With Spliceosome Mutations or Ring Sideroblasts)
All-Cause Mortality (participants affected / at risk) | 13/19 | 15/16 | 9/9 | 8/9 | 9/18 | 6/9
Serious Adverse Events (participants affected / at risk) | 17/19 | 12/16 | 9/9 | 7/9 | 14/18 | 9/9
Other Adverse Events (participants affected / at risk) | 19/19 | 16/16 | 9/9 | 9/9 | 18/18 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Imetelstat 9.4 mg/kg (MF) (N=19) | Arm B: Imetelstat 9.4 mg/kg as Induction + Maintenance (MF) (N=16) | Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia (N=9) | Arm E: Imetelstat 7.5 - 9.4 mg/kg (MF [With Spliceosome Mutation or Ring Sideroblasts]) (N=9) | Arm F: Imetelstat 7.5 - 9.4 mg/kg (MF [Without Spliceosome Mutation and Ring Sideroblasts]) (N=18) | Arm G: Imetelstat 7.5 - 9.4 mg/kg (MDS/MPN or MDS With Spliceosome Mutations or Ring Sideroblasts) (N=9)
Platelet count decreased (Investigations) | 10 | 5 | 8 | 5 | 3 | 1
Neutrophil count decreased (Investigations) | 4 | 6 | 5 | 1 | 3 | 5
White blood cell count decreased (Investigations) | 3 | 6 | 1 | 0 | 4 | 2
Anaemia (Blood and lymphatic system disorders) | 9 | 10 | 8 | 5 | 7 | 8
Lung infection (Infections and infestations) | 0 | 1 | 3 | 1 | 2 | 1
Sepsis (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 2 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | 0 | 2 | 1
Fatigue (General disorders) | 1 | 1 | 2 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Imetelstat 9.4 mg/kg (MF) (N=19) | Arm B: Imetelstat 9.4 mg/kg as Induction + Maintenance (MF) (N=16) | Arm D: Imetelstat 9.4 mg/kg (Blast-phase MF/Acute Myeloid Leukemia (N=9) | Arm E: Imetelstat 7.5 - 9.4 mg/kg (MF [With Spliceosome Mutation or Ring Sideroblasts]) (N=9) | Arm F: Imetelstat 7.5 - 9.4 mg/kg (MF [Without Spliceosome Mutation and Ring Sideroblasts]) (N=18) | Arm G: Imetelstat 7.5 - 9.4 mg/kg (MDS/MPN or MDS With Spliceosome Mutations or Ring Sideroblasts) (N=9)
Anaemia (Blood and lymphatic system disorders) | 16 | 9 | 4 | 6 | 11 | 7
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 1 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1 | 0 | 0 | 2 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 2 | 0 | 3 | 0
Eye disorders (Eye disorders) | 1 | 1 | 1 | 0 | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 1 | 6 | 2 | 6 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 4 | 1 | 1 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 19 | 15 | 8 | 9 | 18 | 9
Nausea (Gastrointestinal disorders) | 8 | 7 | 6 | 1 | 12 | 4
Vomiting (Gastrointestinal disorders) | 7 | 3 | 1 | 1 | 5 | 1
Chills (General disorders) | 3 | 2 | 2 | 1 | 2 | 0
Early satiety (General disorders) | 4 | 3 | 3 | 3 | 1 | 1
Fatigue (General disorders) | 18 | 15 | 8 | 8 | 18 | 9
Infusion related reaction (General disorders) | 2 | 3 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 2 | 0 | 1 | 0 | 1 | 1
Oedema peripheral (General disorders) | 7 | 3 | 6 | 3 | 5 | 2
Pain (General disorders) | 6 | 5 | 3 | 2 | 8 | 5
Pyrexia (General disorders) | 5 | 2 | 4 | 1 | 2 | 1
Lung infection (Infections and infestations) | 1 | 1 | 3 | 1 | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 4 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 3 | 1 | 1 | 3 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 3 | 1
Activated partial thromboplastin time prolonged (Investigations) | 10 | 3 | 5 | 2 | 7 | 0
Alanine aminotransferase increased (Investigations) | 8 | 3 | 4 | 2 | 6 | 5
Aspartate aminotransferase increased (Investigations) | 10 | 8 | 4 | 3 | 6 | 5
Blood alkaline phosphatase increased (Investigations) | 10 | 10 | 3 | 4 | 5 | 1
Blood amylase increased (Investigations) | 3 | 0 | 2 | 1 | 2 | 2
Blood bilirubin increased (Investigations) | 7 | 5 | 1 | 1 | 5 | 3
Blood creatinine increased (Investigations) | 4 | 2 | 4 | 0 | 4 | 4
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 0 | 0 | 4 | 1
Lipase increased (Investigations) | 3 | 1 | 3 | 2 | 3 | 3
Lymphocyte count decreased (Investigations) | 1 | 1 | 0 | 0 | 2 | 1
Neutrophil count decreased (Investigations) | 19 | 16 | 9 | 9 | 18 | 9
Platelet count decreased (Investigations) | 19 | 16 | 9 | 9 | 18 | 9
Weight decreased (Investigations) | 1 | 4 | 0 | 0 | 6 | 2
Weight increased (Investigations) | 1 | 1 | 0 | 0 | 2 | 2
White blood cell count decreased (Investigations) | 19 | 16 | 9 | 9 | 18 | 9
Anorexia (Metabolism and nutrition disorders) | 4 | 5 | 4 | 1 | 4 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 10 | 7 | 4 | 13 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 4 | 2 | 2 | 3 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 2 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 8 | 5 | 2 | 2 | 8 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 2 | 4 | 0 | 3 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 3 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0 | 2 | 0 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2 | 3 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 1 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1 | 1 | 3 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 1 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 3 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3 | 1 | 2 | 2
Dizziness (Nervous system disorders) | 3 | 0 | 3 | 1 | 0 | 1
Headache (Nervous system disorders) | 4 | 2 | 0 | 0 | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 1 | 0 | 2 | 1
Insomnia (Psychiatric disorders) | 3 | 2 | 2 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 4 | 3 | 5 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 7 | 2 | 5 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 1 | 1 | 4 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 0 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 2 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1 | 0 | 1 | 4 | 0
Haematoma (Vascular disorders) | 1 | 2 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 5 | 2
Hypotension (Vascular disorders) | 1 | 0 | 3 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Consistent with Good Publication Practices and ICMJE guidelines, the sponsor shall have right to publish such primary (multicenter) data and information without approval from investigator. Investigator has right to publish study site-specific data after primary data published. If an investigator wishes to publish information from study, a copy of manuscript must be provided to sponsor for review at least 60 days before submission for publication or presentation

DOCUMENTS (2):
  • Study Protocol (2015-10-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT01731951/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT01731951/SAP_001.pdf